CLINICAL TRIAL: NCT01737567
Title: A Randomised Comparison Between White Light Endoscopy (WLE) and Bright Narrow Band Imaging (B-NBI) in the Diagnosis of Colonic Adenomas in Asymptomatic Subjects Undergoing Screening Colonoscopy.
Brief Title: Comparison Between White Light Endoscopy and Bright Narrow Band Imaging in Diagnosis Colonic Adenomas.
Acronym: WLEvB-NBI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: similar study is progressing instead
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HREC/11/WMEAD/223; HREC2011/12/4.9 (3395) (Other: HREC WSLHD)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colonic Adenomas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bright Narrow Band Imaging (Experimental): Use of B-NBI to detect colonic adenomas.
  Interventions: Other: Bright Narrow Band Imaging.
- White Light Endoscopy (Active Comparator): Use of White Light Endoscopy to detect colonic adenomas.
  Interventions: Other: White Light Endoscopy

INTERVENTIONS:
Other: Bright Narrow Band Imaging. — Using Bright Narrow Band Imaging to detect colonic adenomas.
  Arms: Bright Narrow Band Imaging
Other: White Light Endoscopy — Use of White Light Endoscopy to detect colonic adenomas.
  Arms: White Light Endoscopy

SUMMARY:
Removal of colorectal adenomas prevents the occurence of colorectal cancers. The use of chromo-endoscopy has been shown to improve the detection of flat adenomas. Narrow band imaging enables endoscopists to accurately describe the pit pattern of adenomas. By comparing White Light Endoscopy and Bright Narrow Band Imaging it will show if there is any comparable advantage to using one or the other for lesion detection and assessment.

DETAILED DESCRIPTION:
Removal of colorectal adenomas prevents occurrence of cancers [1]. It is recognized that colonoscopy can miss colorectal adenomas and early cancers [2]. There is a need to further improve performance of colonoscopy. The use of chromoendoscopy has been shown to improve detection of flat adenomas [3]. Narrow band imaging was introduced in year 2006. It is similar to chromoendoscopy in that it provides more mucosal details. This enables endoscopists to accurately describe the pit pattern of adenomas. NBI has been used as a substitute to chromoendoscopy.

In pooled analysis, NBI is comparable to chromoendoscopy in their sensitivity and specificity in the diagnosis of malignant colorectal adenomas [4]. Unfortunately, the use of NBI has not been shown to conclusively improve rate of colorectal adenoma detection. Two of 3 randomized trials that compared WLE to NBI showed a higher adenoma detection rate with the use of NBI [5, 6]. In a study by Rex et al., the rate was however similar with either modality. In a pooled analysis, NBI was only marginally better than WLE [7].

The effective use of NBI depends on the quality of bowel preparation and the experience of endoscopist. In the presence of fecal matters, NBI tends to be dark and detection of small adenomas becomes difficult. The prototype bright NBI coupled with high definition resolution is likely to overcome this drawback of original NBI.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects undergoing screening colonoscopy, age > 50, average risk subjects and, ability to provide a written consent to trial participation.

Exclusion Criteria:

* personal history of inflammatory bowel disease, colon adenoma or cancer
* family history of FAP or Familial nonpolyposis syndrome
* first degree relatives having diagnosed to have colorectal carcinoma
* no colonoscopy in past 5 years

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2021-06 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in detection of colorectal adenomas. | One year
  It is anticipated that colorectal adenomas will be more easily identifiable using Bright Narrow Band Imaging.

SECONDARY OUTCOMES:
Improvement of histological prediction | One year
  It is anticipated that the use of Bright Narrow Band Imaging will significantly improve the histological detection of colonic adenomas when detected as opposed to White Light Endoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia